CLINICAL TRIAL: NCT04749381
Title: The Role of Traditional Chinese Medicine on Enhanced Recovery After Surgery for Patients With Rectal Cancer Undergoing Curative Surgery: A Randomized Controlled Trial
Brief Title: The Role of TCM on ERAS of Rectal Cancer Patients
Acronym: RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, M.D. PH.D. Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKUCH-R06
Record Dates: First submitted 2020-10-09; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer
Keywords: ERAS; Integrative medicine; Acupoint application; Compliance; Quality of life
MeSH Terms: conditions — Rectal Neoplasms; Patient Compliance | interventions — Acupuncture Points

STUDY DESIGN:
Intervention Model Description: Patients enrolled are randomized into acupoint application group and placebo acupoint application group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM group (Experimental): Rectal cancer patients randomized to this group will have acupoint application with traditional Chinese medicine.
  Interventions: Combination Product: acupoint with TCM
- Control group (Placebo Comparator): Rectal cancer patients randomized to this group will have acupoint application with placebo .
  Interventions: Combination Product: acupoint with placebo

INTERVENTIONS:
Combination Product: acupoint with TCM — The acupoint application was made of traditional Chinese medicine (TCM), and the therapeutic effect was produced through the stimulation of TCM drugs and acupoints.
  Arms: TCM group
Combination Product: acupoint with placebo — The placebo acupoint application was made of black beans and honey, which shares the similar shape and smell of the experiment group, applied at the same acupoints.
  Arms: Control group

SUMMARY:
This study is to investigate the role of traditional Chinese medicine (TCM) on the postoperative recovery of rectal cancer patients.

DETAILED DESCRIPTION:
The hypothesis is that TCM can decrease the postoperative complications for rectal cancer. So the study is to investigate the role of traditional Chinese medicine (TCM) on the postoperative recovery of rectal cancer patients. Patients enrolled in this study will be randomized into two groups with TCM intervention or placebo. The intervention will be described below. Primary endpoint is postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form;
* Age from 18 to 75 years old;
* Pathological diagnosis as rectal adenocarcinoma;
* undergo laparoscopic curative surgery;
* Patients' TCM syndrome accords with thoses of spleen deficiency syndrome;

Exclusion Criteria:

* Patients undergo non-curative surgeries;
* Participants with skin allergy, skin ulceration and diabetes mellitus with poor glycemic control;
* Participants with severe dysfunction of heart, liver and kidney, who could not receive TCM treatment;
* Women who are pregnant or breastfeeding;
* Participants have mental illness or have difficulty in language communication and are unable to complete the study;
* Participants could not cooperate with this researcher for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | from operation to 30 days after operation
  Rates of the complications after curative surgery

SECONDARY OUTCOMES:
recovery of urinary function | from removal of urinary catheter to 30 days after operation
  The rates of urinary retention after removal of urinary catheter
Recovery of fart and bowel function | 7 days after operation
  The time of the first tart and first defecation after operation in days
The European Organization of Quality of Life Questionnaire-colorectal-29 | 30 days after operation
  Cancer Quality of Life Questionnaire-Colorectal-29, with scale from 1 to 4 for each items as QOL becomes poorer.
Changes of TCM symptoms | 30 days after operation
  Changes of traditional Chinese medicine symptoms: all symptoms were recorded by 10 simple questions and then will be categorized in 4 different groups. The aim of study tries to show the relationship with TCM application with the symptoms.
Length of hospital stay | 30 days after operation
  Time of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute; Xiaoqiang Jia, M.D.;Ph.D, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China